CLINICAL TRIAL: NCT04362449
Title: A Prospective Study of Tolerance Comparing the Current Hydration Regimen for the ABC02 Chemotherapy Regimen Versus a Shorter Hydration
Brief Title: Comparing the Current Hydration Regimen for the ABC02 Chemotherapy Regimen Versus a Shorter Hydration
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Chugai Pharma UK Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 214262
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Gallbladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shortened hydration time with dispensary of Akynzeo (Experimental): ABC-02 regime - gemcitabine and cisplatin with a shortened hydration time and administration of a newer antiemetic
  Interventions: Combination Product: Shortened hydration time and dispensary of Akynzeo
- Standard of care (Active Comparator): ABC-02 regime - gemcitabine and cisplatin with currently approved hydration time and administration of the current choice of antiemetic
  Interventions: Combination Product: Standard of care

INTERVENTIONS:
Combination Product: Shortened hydration time and dispensary of Akynzeo — Hydration is reduced to 1 hour and 40 minutes and Akynzeo is administered as an oral drug instead of Ondansetron being given as an IV before chemotherapy.
  Arms: Shortened hydration time with dispensary of Akynzeo
Combination Product: Standard of care — Hydration remains at around 6 hours and 30 minutes due to no oral fluids being consumed prior to treatment and normal saline being administered for 90 minutes before cisplatin and then for 2 hours after cisplatin and before gemcitabine administration
  Arms: Standard of care

SUMMARY:
This is an open label study for any patients with a bile duct cancer or gallbladder cancer, who will be treated with gemcitabine and cisplatin chemotherapy (the ABC02 regime). Patients recruited onto this study will have a reduction of their hydration time and be given Akynzeo as an anti-sickness drug, to assess tolerability compared to the current standard of care. The aim of this research is to assess the tolerability of a shorter hydration time, which may improve patient satisfaction as they would then spend less time in hospital having chemotherapy, saving both time and money for the institutions also.

DETAILED DESCRIPTION:
The ABC02 treatment regime was established in 2010 following publication in the New England Journal of Medicine and has since become the standard of care treatment of bile duct cancers otherwise known as cholangiocarcinomas, as well as gallbladder cancer. The treatment consists of gemcitabine and cisplatin given synergistically. This combination has been shown to yield an overall survival advantage of 3.6 months compared to when gemcitabine is given on its own, with additional improvements in performance status and tumour control in patients.

Currently, the ABC02 regime includes a long hydration schedule based on previous use of high doses of cisplatin and perhaps historically the lack of efficacious antiemetics. Cisplatin is often associated with severe nausea and vomiting that lead to dehydration. In fact, cisplatin is a direct nephrotoxin, owing to its pro-inflammatory action in the kidneys and being able to cause immediate vasoconstriction of renal microvasculature on administration, and this coupled with its effect to induce dehydration due to nausea and vomiting, prevented the inclusion of cisplatin into many combinational regimens. 50% of patients in initial studies were found to suffer from nephrotoxicity on cisplatin and thus the administration of intravenous saline to combat this effect by inducing diuresis has also been standard of care when giving cisplatin chemotherapy. However, it is still not known what the optimal hydration solution and procedure are as there are no studies comparing either of these factors.

Akynzeo is a mixture of both a 5HT3 blocker palonosetron and a neurokinin 1 inhibitor netupitant. Together the drugs are able to combat nausea and vomiting during the acute phase and delayed phase after chemotherapy. The introduction of 5HT3 blockers cut the incidence of acute nausea and vomiting in chemotherapy patients considerably, but in fear of the historical nephrotoxicity, copious volumes of IV saline remains part of the regime. This entire procedure takes 8 hours for delivery and risks fluid overload often requiring diuretic management.

For reference: gemcitabine is an antimetabolite and works by imitating a pyrimidine and replacing the cytidine in nucleic acid during DNA replication. By doing so, gemcitabine halts tumour growth as actual nucleosides cannot be attached to this faulty nucleoside and this results in apoptosis. Cisplatin on the other hand is an alkylating agent and kills cancer cells by binding to DNA and interfering with its repair mechanism; upon binding to DNA it further attracts other DNA repair proteins to irreversibly bind to the structure distorting its shape and inducing apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults with normal renal function at the start i.e. eGFR>60, Performance status 0 and 1, controlled nausea and vomiting at baseline.
* ECOG performance status 0 or 1
* Diagnosed with either cholangio carcinoma, gallbladder cancer, pulmonary cancer or pancreatic cancer. Patients should be able to tolerate 1 litre of oral fluid pre-treatment and post treatment.
* Decision to treat with the gemcitabine and cisplatin used in the ABC02 trial.

Exclusion Criteria:

* Participants under the age of 18 years old with Chronic renal impairment. The standard exclusion of renal impairment for cisplatin implies that this study would not be offered to patients, who can't be safely offered cisplatin
* Uncontrolled nausea or vomiting
* Unable to drink 1 litre of fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-02-02 (Estimated); Study Completion 2023-02-02 (Estimated)

PRIMARY OUTCOMES:
Nausea according to the Common Terminology Criteria for Adverse Events (CTCAE) V4.03 | Throughout study completion, up to 1 year
  To compare the proportion of patients who experience CTCAE V3.0 grade 3 or 4 nausea (using a shortened hydration protocol and a modern antiemetic regimen) with those who are in the ABC02 trial arm which used a longer hydration procedure and a standard antiemetic regimen

SECONDARY OUTCOMES:
Renal function of patients | Throughout study completion, up to 1 year
  To compare proportion of patients who experience CTCAE V3.0 grade 3 or 4 impaired renal function
Number of patients who have a complete response | Throughout study completion, up to 1 year
  To compare proportion of patients who have a complete response i.e. no nausea and vomiting recorded as a toxicity
Number of patients with renal dysfunction | Throughout study completion, up to 1 year
  To compare the proportion of patients who experience renal dysfunction (a deterioration of calculated GFR of below 60)
Number of cases of chemotherapy induced emesis | Throughout study completion, up to 1 year
  To determine the incidence of early and delayed chemotherapy induced emesis using the MAT antiemesis tool
Nocturia experienced by patients | Throughout study completion, up to 1 year
  To determine the incidence of nocturia in the first night after chemotherapy
Health economics in the context of duration of hospital attendance | Throughout study completion, up to 1 year
  Measuring the length of hospital visit (time in to time out) for each patient per treatment visit and comparing the difference between arms

CONTACTS AND LOCATIONS:
Overall Officials: Harpreet Wasan, MD, Principal Investigator — Gastrointestinal Clinical Research Lead and Consultant Oncologist
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided